CLINICAL TRIAL: NCT05151770
Title: Type 1 Diabetic Post Prandial Glycemia Evaluation Using an Algorithm
Acronym: EGHYA
Status: Completed | Type: Observational
Sponsor: M-DT1 (Industry)
Collaborators: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other); Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-MDT1-001; 2021-AO2599-32 (Other: Centre intercommunal Toulon La seine sur Mer)
Record Dates: First submitted 2021-11-12; First posted 2021-12-09 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2022-04

CONDITIONS: Type I Diabetes
Keywords: Type I diabetes; Hyperglycemia; Post prandial glycemia; algorithm
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hyperglycemia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measure of glycemia levels and comparison to algorithm predictions — The study aims to evaluate the efficacy of a new algorithm in predicting the evolution of glycemia levels after a full meal. Glycemia levels measured during and after a full meal will be compared to the values predicted by the algorithm. Composition of the meals will also be collected.

SUMMARY:
The aim of this study is to demonstrate the efficacy of an algorithm to anticipate the post prandial glycemic profile in type I diabetic patient.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* ≥ 18 years old
* Hb1Ac<12%

Exclusion Criteria:

* Patient without continuous glucose monitoring system
* Disease other than diabetes (bulimia, anorexia…)
* Dialysis patient
* Known history of drug or alcohol abuse
* Patient under judicial protection
* Person deprived of liberty
* Pregnant, parturient or breastfeeding woman
* Patient in psychiatric care
* Patient admitted to a health or social institution for purposes other than research
* Any reasons that might interfere with the evaluation of the study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type I diabetes
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2021-12-30 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Algorithm efficacy | 15 days
  The Algorithm efficacy in predicting the risk or absence of risk of hyperglycemia two hours after taking a full meal is evaluated by comparing glycemic values calculated by the algorithm and those obtained using continuous glucose monitoring system measurements.

SECONDARY OUTCOMES:
Algorithm efficacy (lower margin of error) | 15 days
  The Algorithm efficacy in predicting the risk or absence of risk of hyperglycemia two hours after taking a full meal is evaluated by comparing glycemic values calculated by the algorithm and those obtained using continuous glucose monitoring system measurements (the accepted margin of error is reduced by 25 to 50% when compared with primary outcome).
Algorithm efficacy versus meal composition | 15 days
  Meals will be analyzed within different groups according to their respective nutritional index. For each group, algorithm prediction reliability will be determined.
Influence of the age of the patients on algorithm results | 15 days
  The Algorithm efficacy will be analyzed according to the age of patients
Influence of the BMI on algorithms results | 15 days
  Weight and height of patients will be combined to report BMI in kg/m2. Algorithm efficacy will be analyzed according to the BMI of patients
Influence of the insulin administration on algorithm results | 15 days
  Data obtained from patients using insulin pumps will be compared to data obtained from patients using multiple daily insulin injections.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - APHM, Marseille
  - Hopital Sainte Musse, Toulon

IPD SHARING:
Plan to Share IPD: No